CLINICAL TRIAL: NCT05349734
Title: Comparison of Upper Body and Full Underbody Forced Air Blanket for Maintaining Normothermia in Pediatric Patients Undergoing Cardiovascular Interventions Under General Anesthesia: a Randomized Controlled Trial
Brief Title: Comparison of Upper Body and Full Underbody Forced Air Blanket in Pediatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hee-Soo Kim, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2005-016-1121
Record Dates: First submitted 2022-04-09; First posted 2022-04-27 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Hypothermia; Anesthesia
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- upper body (Experimental)
  Interventions: Other: upper body blanket
- full underbody (Active Comparator)
  Interventions: Other: full underbody blanket

INTERVENTIONS:
Other: upper body blanket — applying upper body blanket with forced-air blower set to 43℃
  Arms: upper body
Other: full underbody blanket — applying full underbody blanket with forced-air blower set to 43℃
  Arms: full underbody

SUMMARY:
The aim of this study is to compare the underbody blanket and overbody blanket for forced air warming to maintain normothermia in pediatric patients undergoing cardiovascular interventions under general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* pediatric patients under 15 years of age who are scheduled for cardiovascular interventions in angioroom

Exclusion Criteria:

* anticipated operating time < 1 hour
* body surface area that exposured by drape < 30% of total body surface area
* BMI > 30
* corrected age < 40 weeks
* preoperative body temperature is higher than 37℃ or less than 35.5℃
* patients with skin disease
* history of malignant hyperthermia
* patients who cannot use esophageal stethoscope

Ages: 1 Day to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 92 (Actual)
Dates: Start 2022-05-12 (Actual); Primary Completion 2023-03-02 (Actual); Study Completion 2023-03-03 (Actual)

PRIMARY OUTCOMES:
hypothermia | intraoperative period (from the time when patient enters the operating room to the time when patient exits the operating room)
  time weighted average out of normothernia (body temperature over 37.5℃ and under 36.5℃) in intraoperative period

SECONDARY OUTCOMES:
hyperthermia | intraoperative period (from the time when patient enters the operating room to the time when patient exits the operating room)
  body temperature recorded over 37.5℃
thermal comfort scale | 15 minutes, 30 minutes, 45 minutes, 60 minutes after entering the post-anesthesia care unit
  asking subjects about the thermal sensation on a seven-point scale from cold(-3) to hot (+3)
patient satifisfaction at post-anesthesia care unit | 15 minutes, 30 minutes, 45 minutes, 60 minutes after entering the post-anesthesia care unit
  visual analog scale score for measuring the patient satisfaction after the surgery (0~10)
shivering score at post-anesthesia care unit | 15 minutes, 30 minutes, 45 minutes, 60 minutes after entering the post-anesthesia care unit
  4 grades of shivering score measured at post-anesthesia care unit
clinical outcomes after the surgery | 5 days after the surgery
  postoperative complications during hospitalization

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Park JB, Kim TW, Ji SH, Jang YE, Lee JH, Kim JT, Kim HS, Kim EH. Comparison between upper body and full underbody forced-air warming blanket in pediatric patients undergoing cardiovascular interventions under general anesthesia: a randomized controlled trial. BMC Anesthesiol. 2025 May 21;25(1):254. doi: 10.1186/s12871-025-03100-3. PMID 40399788